CLINICAL TRIAL: NCT02050152
Title: Dose Response Effect of Nitrous Oxide on Amnesia in Healthy Children
Brief Title: Nitrous Oxide Induction Induces Amnesia in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jerrold Lerman, Clinical Professor of Anesthesiology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Nitrous Oxide Amnesia Children
Record Dates: First submitted 2013-03-22; First posted 2014-01-30 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Amnesia
Keywords: Amnesia; Memory; Implicit; Explicit; Nitrous Oxide
MeSH Terms: conditions — Amnesia | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0% nitrous oxide (Placebo Comparator): Explicit and implicit memory will be tested in 0% nitrous oxide
  Interventions: Behavioral: Explicit and Implicit memory; Drug: 0% nitrous oxide, 30% nitrous oxide and 60% nitrous oxide
- 30% nitrous oxide (Active Comparator): Explicit and Implicit memory in 30% nitrous oxide
  Interventions: Behavioral: Explicit and Implicit memory; Drug: 0% nitrous oxide, 30% nitrous oxide and 60% nitrous oxide
- 60% nitrous oxide (Active Comparator): Explicit and Implicit memory with 60% nitrous oxide
  Interventions: Behavioral: Explicit and Implicit memory; Drug: 0% nitrous oxide, 30% nitrous oxide and 60% nitrous oxide

INTERVENTIONS:
Behavioral: Explicit and Implicit memory — Explicit and implicit memory will be tested visually (showing an animal) and auditory (telling a joke, stating a food type that starts with the letter B) and smell recall (bad smell of anesthesia)
Drug: 0% nitrous oxide, 30% nitrous oxide and 60% nitrous oxide

SUMMARY:
The investigators are conducting a study to investigate the amnestic effects of 2 different concentrations of nitrous oxide in children before induction of anesthesia in a prospective double-blinded placebo controlled study.

DETAILED DESCRIPTION:
Children of age group 6-12 will be randomly divided in 3 groups, First group will be Placebo , second group will be nitrous oxide end tidal 20-30% and third group will be nitrous oxide 60-70%. Each group will be divided into 2 subgroups randomly with either a flavored or unflavored mask for induction.

All children will be told a joke before the mask is applied, with the answer provided after the end-tidal nitrous oxide concentration reaches the randomized concentration (0, 30 or 60%) for at least one minute. At that point, the child will randomized to be either shown a picture of one of four animals (predetermined randomly) or a food will be stated aloud. For the animal, the child will be asked to name the animal aloud. The child's response (yes or no to a response and whether the item is correctly named) will be recorded. If the child does not respond, the name of the animal will be stated out loud. For the food, one of four foods will be named aloud and child will be asked to repeat the name. The child's response (named or not) will be recorded. Anesthesia will continue with the designated nitrous oxide concentration combined with 8% Sevoflurane.

When the child is ready for discharge from the recovery room and recovered from anesthesia, a nurse or doctor who is blinded to the treatment group assignment will ask the child to recall the joke and answer. The child will then be asked if they were shown any animals and if so, which animal? If the child cannot recall an animal, the child will be asked to name the first animal that comes to mind. The child will then be shown pictures of four animals and asked to identify one. The child will be asked if they heard any foods when they went to sleep? If the child cannot recall hearing any foods recited, the first letter of the food will be shown: B _ _ _ _ _ . If the child does not recall any foods, then the child will be given the names of four foods that begin with the letter B and asked to pick one. Finally, the child will be asked about any odors in the mask during anesthesia. If he/she does not recall, then four odors will be read out and the child asked to identify any one. Additionally, the children will be asked whether they recall any odors on the mask as they were anesthetized. The order of items questioned in the recovery period will follow the same order as in the OR.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6-12 years old,
2. ASA classification: 1 and 2
3. Elective surgery

Exclusion Criteria:

1. Uncooperative child needs sedation before induction of anesthesia
2. Developmental delay, ADHD, autism, Tourette's syndrome, schizophrenia, congenital and acquired brain disorder, Down syndrome.
3. Those who request for IV induction
4. Those taking sedative medications, anti-seizure medication
5. Those with malignant hyperthermia, muscular dystrophy; those with uncorrected cardiac defects and those with severe or active lung disease
6. Those with elective admissions to PICU with ongoing sedation and tracheal intubation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Nitrous Oxide effects on explicit memory | After full recovery from anesthesia (generally by 2 hours after termination of anesthesia), but before discharge from hospital all variables will be assessed
  Explicit and implicit memory will be tested during the recovery period (once the child has fully recovered from anesthesia but before discharge from hospital) by a blinded observer who will ask the child to recall the joke they were told, the animal picture they were shown, the name of the food they heard and any odor they noticed as they fell asleep

SECONDARY OUTCOMES:
Nitrous oxide effect on Implicit memory | After recovery from anesthesia (in recovery room or before discharge from hospital) within 4 hours of anesthesia completion
  Implicit memory will be tested if the child fails to identify any of the explicit tests by showing the child four animal pictures and picking an animal or by reciting four foods and asking the child to pick one.

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Lerman, MD, FRCPC, Principal Investigator — Professor
Locations (1):
- Women and Children's Hospital of Buffalo, Buffalo, New York, United States